CLINICAL TRIAL: NCT00720265
Title: A PHASE III, Randomized, Open-Label, Comparative, Multi - Center Study to Assess the Safety and Efficacy of Prograf® (Tacrolimus) and MR4 (Modified Release Tacrolimus) in de Novo Kidney Transplant Recipients
Brief Title: A Study to Assess the Safety and Efficacy of Prograf and MR4 in Kidney Transplantation Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-05-01-KOR
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Kidney Transplantation
Keywords: Organ Transplantation; Tacrolimus; Prograf; FK506MR
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Prograf
- 2 (Experimental)
  Interventions: Drug: MR4

INTERVENTIONS:
Drug: Prograf — oral
  Other Names: Tacrolimus; FK506
  Arms: 1
Drug: MR4 — oral
  Other Names: Modified Release Tacrolimus; FK506MR; FK506E
  Arms: 2

SUMMARY:
To prove non-inferiority of MR4 to Prograf by evaluating the efficacy and safety of Prograf and MR4 in new kidney transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Patient must receive first oral dose of randomized study drug 2days(min 1day) prior to transplant procedure
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within 7 days prior to enrollment

Exclusion Criteria:

* Patient has previously received an organ transplant other than a kidney
* Patient has received a Kidney transplant from non-heart beating donor or a cadaveric donor
* Patients has received an ABO incompatible donor kidney
* Recipient or donor is known to be seropositive for human immunodeficiency virus(HIV)
* Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Patient has significant liver, disease, defined as having during the past 28 days continuously elevated AST (SGOT) and/or ALT (SGPT) levels greater than 3 times the upper value of the normal range of the investigational site
* Patient has an uncontrolled concomitant infection(including Hepatitis B, Hepatitis C)or any other unstable medical condition that could interfere with the study objectives
* Patient is currently taking or has been taking an immunosuppressive agents in the 30 days prior to transplant(except from two days prior to transplant)
* Patient has a known hypersensitivity to tacrolimus
* Patient is pregnant or lactating

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Acute rejection within 24 weeks (6 months) | 6 months

SECONDARY OUTCOMES:
Incidence of biopsy-proven acute rejection (Banff Grade ≥ 1) | at 6 months
Time to first acute rejection episode | for 6 months
6 month patient and graft survival rate | at 6 months
Severity of acute rejection | 6 months
Adverse events, laboratory parameters and vital signs | Throughout trial

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Korea, Inc.
Locations (2):
- South Korea (2):
  - Daegu
  - Seoul